CLINICAL TRIAL: NCT03969550
Title: Do CCR5 Antagonists Improve the Overall Survival of Patients With AIDS-related Progressive Multifocal Leucoencephalopathy?
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: 29305436
Record Dates: First submitted 2019-05-29; First posted 2019-05-31 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: AIDS; Progressive Multifocal Leucoencephalopathy (PML)
Keywords: Maraviroc; John Cunningham virus (JCV); Immune reconstitution inflammatory syndrome (IRIS); Combined antiretroviral treatment (cART); Overall survival (OS)
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Leukoencephalopathy, Progressive Multifocal; Immune Reconstitution Inflammatory Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Measure of overall survival — Measure of overall survival among AR-PML (AIDS-related PML) patients, exposed or not to maraviroc (MVC), and immune reconstitution inflammatory syndrome (IRIS) onset.

SUMMARY:
Progressive multifocal leucoencephalopathy (PML) is a demyelinating disease caused by John Cunningham virus (JCV) reactivation. Numerous molecules have been overstated because there were inaccurately tested in non-rigorous clinical trial.

The objective is to draw lessons from repeatedly false hopes of unconfirmed PML treatments that might contribute to prescribing ineffective drugs on claimed efficacy in case reports or small series and by failing to respect the need for clinical trial evaluation before authorizing their widespread use.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AR-PML
* Diagnosed between January 2008 and December 2015
* Followed in one of the four University Hospitals' Infectious Diseases Departments

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with AR-PML, exposed or not to maraviroc, as part of combined antiretroviral treatment (cART).
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | 8 years

IPD SHARING:
Plan to Share IPD: No